CLINICAL TRIAL: NCT05871866
Title: The Use of a Minimally Invasive Internal Fixation Device for Treatment of Unstable Pelvic Ring Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Essam Ahmed, Assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-23-04-01MD
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Unstable Pelvic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: minimally invasive internal fixation device "infix" — An INFIX involves the insertion of spinal pedicle screws in the anterior pelvis (supra-acetabular entry) and the placement of a connecting rod in the subcutaneous tissue of the patient

SUMMARY:
Pelvic fractures are common presentations to major trauma centers and are associated with significant morbidity in polytrauma patients. Traditional open reduction and internal fixation is associated with a high incidence of surgical morbidity, while external fixators, used for both temporary stabilisation and as definitive management, have a complication rate of up to 62% [4], with poor patient tolerance, pin site infection and aseptic loosening the more commonly documented complications in the literature.

Minimally invasive techniques have become more popular recently in the management of pelvic injuries due to their lower incidence of surgical morbidity. The application of a pelvic internal fixator (INFIX) has been presented as a comparable alternative to external fixation of anterior pelvic ring injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had APC-II
* Patients who had APC-III
* Patients who had LC - II
* Patients who had LC -III

Exclusion Criteria:

* Patients who had immature skeletons or medical contraindications such as combined neurovascular injuries and uncontrolled medical diseases.
* Open fractures.
* Stable pelvic ring fractures.
* Patients who had combined acetabular fractures
* Patients who had a hernia or previous lower abdominal surgery.
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
advantages using INFIX | 6 months
  good patient tolerance
union | 1 yea
  radiological

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steer R, Balendra G, Matthews J, Wullschleger M, Reidy J. The use of anterior subcutaneous internal fixation (INFIX) for treatment of pelvic ring injuries in major trauma patients, complications and outcomes. SICOT J. 2019;5:22. doi: 10.1051/sicotj/2019019. Epub 2019 Jun 28. PMID 31250805
- [Background] Lee C, Sciadini M. The Use of External Fixation for the Management of the Unstable Anterior Pelvic Ring. J Orthop Trauma. 2018 Sep;32 Suppl 6:S14-S17. doi: 10.1097/BOT.0000000000001251. PMID 30095676
- [Background] Hoskins W, Bucknill A, Wong J, Britton E, Judson R, Gumm K, Santos R, Sheehy R, Griffin X. A prospective case series for a minimally invasive internal fixation device for anterior pelvic ring fractures. J Orthop Surg Res. 2016 Nov 8;11(1):135. doi: 10.1186/s13018-016-0468-9. PMID 27825365
- [Background] Muller FJ, Stosiek W, Zellner M, Neugebauer R, Fuchtmeier B. The anterior subcutaneous internal fixator (ASIF) for unstable pelvic ring fractures: clinical and radiological mid-term results. Int Orthop. 2013 Nov;37(11):2239-45. doi: 10.1007/s00264-013-2032-0. Epub 2013 Aug 31. PMID 23995332